CLINICAL TRIAL: NCT00562900
Title: Robotic Assisted Versus Laparoscopic Cholecystectomy -
Brief Title: Robotic Assisted Versus Laparoscopic Cholecystectomy - Outcome and Cost Analyses of a Case-Matched Control Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrS_10-07; BrS_10-07
Record Dates: First submitted 2007-11-07; First posted 2007-11-26 (Estimated); Last update posted 2007-11-26 (Estimated); Status verified 2007-11

CONDITIONS: Cholecystolithiasis
MeSH Terms: conditions — Cholecystolithiasis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, robotic (Active Comparator)
  Interventions: Procedure: robotic assisted cholecystectomy
- B, laparoscopic (Active Comparator)
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: robotic assisted cholecystectomy — robotic assisted cholecystectomy
  Arms: A, robotic
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy
  Arms: B, laparoscopic

SUMMARY:
Case matched study on 50 consecutive patients undergoing robotic assisted cholecystectomy (Da Vinci Robot, Intuitive Surgical). These patients are matched 1:1 to 50 patients with conventional laparoscopic cholecystectomy, according to age, gender, ASA score, histology and surgical experience.

* Trial with surgical intervention

DETAILED DESCRIPTION:
Cholecystectomy is used as a starting procedure for robotic-assisted technology in general surgery by most centers. Surprisingly, data is lacking regarding patient outcome or associated costs compared to the use of conventional laparoscopic surgery.

The study is designed to assess the potential benefits of robotic-assisted cholecystectomy. To achieve a high level of evidence we chose a prospective case matched controlled methodology. Three experienced and one junior (2nd yr) surgeon are involved, and were fully trained with the robot prior to initiating the study including tasks in a training box on pig livers and 5 cholecystectomies performed on humans with this technology. Each patient operated with the robotic system is retrospectively matched one by one with patients who underwent a laparoscopic cholecystectomy.

The robotic assisted operations are performed with the 3- arm Da Vinci robot system (Da Vinci Robot, Intuitive Surgical). Similar to the laparoscopic technique an additional fourth trocar was used to retract the gallbladder. The positioning (French) of the patients and the trocars are also comparable to the conventional laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion criteria:

* Cholecystectomy due to symptomatic cholecystolithiasis
* Acute or chronic cholecystitis

Exclusion criteria:

* Patients < 18 years
* Primary open cholecystectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
complications | Dec 04 - Feb 06

SECONDARY OUTCOMES:
Conversion rates, operative time, hospital-costs | Dec 2004 - Feb 2006

CONTACTS AND LOCATIONS:
Overall Officials: stefan breitenstein, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Breitenstein S, Nocito A, Puhan M, Held U, Weber M, Clavien PA. Robotic-assisted versus laparoscopic cholecystectomy: outcome and cost analyses of a case-matched control study. Ann Surg. 2008 Jun;247(6):987-93. doi: 10.1097/SLA.0b013e318172501f. PMID 18520226